CLINICAL TRIAL: NCT07223541
Title: A Randomized Phase II Trial of Cemiplimab or Cemiplimab and Fianlimab After Stereotactic Body Radiotherapy in Oligo-Metastatic Clear Cell Renal Cell Carcinoma
Brief Title: Cemiplimab or Cemiplimab and Fianlimab After Stereotactic Body Radiotherapy in Clear Cell Renal Cell Carcinoma
Acronym: LAG-BOOST
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-LAG-BOOST
Record Dates: First submitted 2025-10-29; First posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: Stereotactic body radiation therapy (SBRT); Oligo metastatic; ctDNA
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cemiplimab + Fianlimab (Experimental): Cemiplimab, 350 mg, IV, and Fianlimab 1600 mg, IV, q3w for 1 year.
  Patients will undergo treatment with the study drug(s) every 3 weeks for a maximum of 17 cycles (approximately 12 months) or until disease recurrence, unacceptable toxic effects, or intercurrent illness preventing further administration.
  Interventions: Drug: Cemiplimab 350 MG Intravenous Solution; Drug: Fianlimab 1600 MG Intravenous Solution
- Cemiplimab (Active Comparator): Cemiplimab 350 mg, IV, Q3W for 1 year.
  Patients will undergo treatment with the study drug(s) every 3 weeks for a maximum of 17 cycles (approximately 12 months) or until disease recurrence, unacceptable toxic effects, or intercurrent illness preventing further administration.
  Interventions: Drug: Cemiplimab 350 MG Intravenous Solution

INTERVENTIONS:
Drug: Cemiplimab 350 MG Intravenous Solution — Cemiplimab is a fully human monoclonal antibody targeting the immune checkpoint receptor PD-1 on T cells and was invented using Regeneron's proprietary Veloc Immune® technology. By binding to PD-1, cemiplimab (Libtayo) has been shown to block cancer cells from using the PD-1 pathway to suppress T-cell activation.
  Other Names: Libtayo
Drug: Fianlimab 1600 MG Intravenous Solution — Fianlimab is a recombinant fully human monoclonal antibody (based on IgG4 isotype) targeting the immune checkpoint receptor LAG-3 on T cells and was invented using Regeneron's proprietary Veloc Immune® technology.
  Arms: Cemiplimab + Fianlimab

SUMMARY:
The purpose of this research is to test the safety of PD-1 inhibitor cemiplimab with or without LAG-3 inhibitor fianlimab, and see what effects (good and bad) of cemiplimab either alone or combined with fianlimab has on patients with oligometastatic clear cell renal cell carcinoma after completion of radiation therapy.

DETAILED DESCRIPTION:
All eligible patients will undergo standard of care SBRT to primary tumor (if present) and/or all metastatic tumor sites prior to randomization. During radiotherapy, patients will receive 1 to 5 fractions delivered over 1-2 weeks.

Then patients will be randomized at 1:1 ratio to the two arms:

* ARM A: Cemiplimab, 350 mg, IV, and Fianlimab 1600 mg, IV, q3w for 1 year,
* ARM B: Cemiplimab 350 mg, IV, Q3W for 1 year. Immune check point inhibition will occur within 3 weeks (+/-1 week) of completion of SBRT

Patients will undergo treatment with the study drug(s) every 3 weeks for a maximum of 17 cycles (approximately 12 months) or until disease recurrence, unacceptable toxic effects, or intercurrent illness preventing further administration.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be >= 18 years of age.
* Patient must have a biopsy/pathologically (histologically or cytologically) proven diagnosis of clear cell renal cell carcinoma (ccRCC) prior to randomization.
* Patient must have at least 1 and not more than 5 metastatic lesions measurable by RECIST v1.1, with imaging obtained within 45 days prior to randomization.
* Patients with untreated brain metastasis measuring <2cm in diameter (intracranial RANO-BM measurable disease required) and with minimal neurological symptoms. Patients with treated brain metastasis are eligible for the trial as long as they have had three or fewer brain metastasis without signs of progression of disease on post-treatment MRI of the brain as per RANO for Brain Metastases (RANO-BM) guidelines.
* Patient must have documentation from a radiation oncologist confirming that all sites (metastases and primary tumor, if present) are amenable to stereotactic body radiation therapy (SBRT).
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* All patients of childbearing potential must have a serum test within 14 days prior to randomization to rule out pregnancy.
* Patient must have the ability to understand and the willingness to sign a written informed consent document.
* Patient must have an Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
* Patients must have adequate organ and bone marrow function per protocol.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial. Testing for HIV is not required for entry onto the study.
* For patients with history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. If no previous history, testing for HBV is not required for entry onto the study.
* For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load. If no previous history, testing for HCV is not required for entry onto the study.
* Patients with prior radiation to sites but without evidence of progression will be allowed, however these RT-treated sites will not be treated on study. Patients who have had a prior nephrectomy can be included in the study, patients with prior metastasectomy are also eligible for the study.

Exclusion Criteria:

* Patients with untreated brain metastasis >2cm, significant neurological deficits and unamenable to surgical resection.
* Patient with variant histology renal cell carcinoma.
* Patient with metastasis invading gastrointestinal tract (such as esophagus, stomach, intestines, colon, rectum).
* Patients with more than 2 liver metastatic lesions, or liver lesions resulting in obstructive jaundice.
* Patient who have received any prior combination systemic therapy for metastatic RCC (including immune checkpoint inhibitors, tyrosine kinase inhibitors or combinations)
* Patients who have received any check point inhibitor or immune therapies (i.e. Vaccine or other immune-oncology agent) within the last 12 months. Patients who have previously been treated for non-metastatic RCC with adjuvant pembrolizumab can be included if over 12 months since last dose and they have not had radiographic progression within 12 months from the last dose of pembrolizumab
* Patients with active autoimmune disease requiring ongoing therapy including systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications daily. Inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Patients with no more than 1 prior systemic therapy for metastatic disease.
* Patients with active tuberculosis per protocol.
* Patients with uncontrolled hypertension (systolic blood pressure [BP] > 190mmHg or diastolic BP > 110mmHg).
* Patients requiring major surgery within 30 days prior to randomization.
* Patients with any serious (requiring hospital stay or long-term rehab) non-healing wound, ulcer, or bone fracture within 30 days prior to randomization.
* Patients with any arterial thrombotic (ST elevation myocardial infarction [STEMI], non-STEMI [NSTEMI], cerebrovascular accident [CVA], etc.) events within 180 days prior to randomization.
* Patients with moderate or severe hepatic impairment (child-Pugh B or C).
* Patients with untreated pulmonary embolism (PE) or deep-vein thrombosis (DVT) is not allowed.
* Patients with unstable cardiac arrhythmia within 180 days prior to randomization.
* Patients with history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, bowel obstruction, or gastric outlet obstruction within 180 days prior to randomization.
* Patients with history of or active inflammatory bowel disease.
* Patients with history of connective tissue disease or other disease in which radiation therapy is contraindicated.
* Patient pregnant or breastfeeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used.
* Patients must not expect to conceive or father children and should use accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study and for 6 months after the last dose of protocol treatment.
* Patients with a history of myocarditis.
* Patients with troponin T (TnT) or troponin I (TnI) > 2x institutional ULN at baseline per protocol.
* Patients with history or current evidence of significant (CTCAE grade ≥2) local or systemic infection (e.g., cellulitis, pneumonia, septicemia) requiring systemic antibiotic treatment within 2 weeks prior to the first dose of trial medication.
* Patients with active infection requiring therapy.
* Patients with ongoing or recent (within 2 years) evidence of an autoimmune disease that required systemic treatment with immunosuppressive agents. The following are non-exclusionary: vitiligo, childhood asthma that has resolved, residual hypothyroidism that requires only hormone replacement, psoriasis not requiring systemic treatment.
* Patients with uncontrolled infection with HIV, HBV, or HCV infection; or diagnosis of immunodeficiency that is related to, or results in chronic infection per protocol.
* Patients with known hypersensitivity to the active substances or to any of the excipients.
* Patients who received a live vaccine within 30 days of planned start of study medication per protocol.
* Women who are fertile following menarche until becoming postmenopausal or women of childbearing potential (WOCBP*), unless permanently sterile must have a negative serum (beta-hCG) at screening per protocol.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with progression-free survival of oligo-metastatic clear cell renal cell carcinoma (ccRCC) patients following stereotactic body radiation therapy (SBRT) and up to one-year of treatment with cemiplimab or cemiplimab plus fianlimab. | 1 year
  Comparison of the 1-year progression-free survival between patients with oligo-metastatic ccRCC treated with cemiplimab alone versus those treated with both cemiplimab and fianlimab following SBRT.

SECONDARY OUTCOMES:
Proportion of TRAEs for assessment of the overall safety profile of cemiplimab and fianlimab in patients with oligo-metastatic ccRCC. | 1 year
  Frequency and severity of TRAEs (Treatment Related Adverse Events), TEAEs (Treatment-Emergent Adverse Events), imAEs (immune-mediated Adverse Events) and SAEs (Severe Adverse Events) related to cemiplimab alone and of cemiplimab + fianlimab by using Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria
Evaluation of the objective response rate (ORR) of cemiplimab and fianlimab | 1 year
  Proportion of patients achieving complete response (CR) or partial response (PR) according to RECIST v1.1 criteria and Response Assessment in Neuro-Oncology (RANO)
Evaluation of the rates of local disease control in patients in response to SBRT with cemiplimab and fianlimab | 1 year
  Proportion of patients with a response rate measurement of time to local progression, measured as per iRECIST guidelines until the date of local progression for each lesion, with death considered a censoring event
Evaluation of the rates of distant disease control in patients in response to SBRT with cemiplimab and fianlimab | 1 year
  Proportion of patients with a response rate measurement of distant progression-free survival (DPFS), measured to the date of first distant progression at a site not documented at registration, or the date of death from any cause for patients without distant progression
Evaluation of duration of response in patients in response to SBRT with cemiplimab and fianlimab | 1 year
  Proportion of patients with a response rate measurement of duration of response (DOR), defined as the time from first documented response (CR or PR) to disease progression or death from any cause
Evaluation of the Overall survival (OS) rate in patients in response to SBRT with cemiplimab and fianlimab | 1 year
  Proportion of patients with a response rate measurement defined as time of enrollment to death from any cause
Evaluation of the rates of disease control in patients in response to SBRT with cemiplimab and fianlimab | 1 year
  Proportion of patients achieving CR, PR, or stable disease (SD) from start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Adanma Ayanambakkam, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States